CLINICAL TRIAL: NCT06805591
Title: Clinical and Imaging Characteristics in Patients Suspected of Dural Leakage Before and After Treatment
Brief Title: Pathophysiology and Treatment of Cerebrospinal Hypotension Exploration Study
Acronym: PATCHES
Status: Enrolling by invitation | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Henrik Schytz, Associate Professor, Consultant Neurologist, Danish Headache Center
Other Study IDs: H-24055595; NNF24OC0087919 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Spontaneous Intracranial Hypotension; Intracranial Hypotension; Post-Lumbar Puncture Headache
Keywords: Spontaneous Intracranial Hypotension; SIH; Post-Lumbar Puncture Headache; PLPH; Danish Headache Center; Post-Dural Puncture Headache; PDPH
MeSH Terms: conditions — Intracranial Hypotension; Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with suspected Intracranial Hypotension: Patients will be included in the cohort if suspected of intracranial hypotension. The group will therefore be subgrouped into patients with spontaneous intracranial Hypotension, post-lumbar puncture headache, and patients suspected but not demonstrated with intracranial hypotension.
- Control Group: Group consisting of healthy control participants.

SUMMARY:
The goal of this observational study is to learn about the effects of a low-pressure environment on the brain in patients with intracranial hypotension and to potentially improve diagnostics and treatment of this condition.

The primary objective will be:

To investigate the change in clinical biomarkers measured before and after successful treatment.

The secondary objectives will be:

To investigate if clinical biomarkers can predict the outcome of treatment. Participants undergoing standard treatment for intracranial hypotension will undergo additional examinations and surveys and will be followed up for a year for the study.

ELIGIBILITY:
Inclusion Criteria (patients):

* Age 18-80.
* Patients with a suspected intracranial hypotension diagnosis.
* Participants must read and understand the Danish language or have an official interpreter present to be able to understand the work-up and sign the participation consent for the study.

Inclusion Criteria (Control):

* Age 18-80.
* Healthy people who do not suffer from any form of primary headache except infrequent tension-type headache.
* Participants must read and understand the Danish language or have an official interpreter present to be able to sign the participation consent for the study.

Exclusion Criteria (patients):

* Pregnant or breastfeeding females
* Patients in whom the examination cannot be performed due to anatomical reasons such as severe head dysmorphia or severe ophthalmological diseases.
* The patient has a disease, takes medication, or abuses alcohol or drugs that could, in the investigator´s opinion interfere with the assessments of safety, tolerability, or efficacy, or interfere with the conduct or interpretation of the study.
* The patient is, in the investigator´s opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Exclusion Criteria (Control):

* Pregnant or breastfeeding females
* Participants in whom the examination cannot be performed due to anatomical reasons such as severe head dysmorphia or severe ophthalmological diseases.
* The participant has a disease, takes medication, or abuses alcohol or drugs that could, in the investigator´s opinion interfere with the interpretation of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at the Danish Headache Center with suspected intracranial hypotension
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
To investigate the change in clinical biomarkers measured before and after successful treatment. | From enrollment to 1 year post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik W Schytz, MD, Ph.D. DMSc, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided